CLINICAL TRIAL: NCT04845165
Title: Study of Cortisol Metabolism in Familial Partial Lipodystrophy Type 2
Acronym: LIPOCORT
Status: Completed | Type: Observational
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: 2020_50; 2020-A03167-32 (Other: ID-RCB number,ANSM)
Record Dates: First submitted 2021-04-13; First posted 2021-04-14 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Familial Partial Lipodystrophy Type 2
Keywords: Cortisol; Lipodystrophy 3; Hydroxysteroid 11-β dehydrogenase 1 (HSD11B1); Insulin Resistance; Hypertriglyceridemia
MeSH Terms: conditions — Lipodystrophy, Familial Partial; Insulin Resistance; Hypertriglyceridemia | interventions — Biopsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — A 24 hours urine collection; Biopsy of subcutaneous adipose tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with FPL2 genetically confirmed: patients suffering with FPL2 with the R482 codon mutation of the LMNA gene.
  Interventions: Other: Biopsy

INTERVENTIONS:
Other: Biopsy — Biopsy of subcutaneous adipose tissue

SUMMARY:
Familial partial lipodystrophic syndromes are characterized by an increase in visceral adipose tissue and an atrophy of subcutaneous adipose tissue. They are associated with a severe metabolic syndrome especially when linked to the mutation of the R482 codon of the LMNA gene (Familial partial lipodystrophy type 2, FPL2). Data in lipodystrophy induced by antiretroviral therapy of HIV suggests an increase in the activity of 11β-hydroxysteroid dehydrogenase type 1 (11bHSD1). This enzyme reactivates cortisone in cortisol in adipose tissues and liver and has associated to obesity and type 2 diabetes mellitus. Hence, the hypothesis is that in patients suffering from FPL2 with the R482 codon mutation of the LMNA gene, there is an increase in the activity of HSD11B1 which could participate to the metabolic phenotype of the disease.

ELIGIBILITY:
Inclusion Criteria:

* Familia partial lipodystrophy type 2 (FPL2) with the R482 codon mutation of the LMNA gene
* Social insured
* Ability to give consent

Exclusion Criteria:

* urinary incontinence or inability to collect urine for 24 hours
* moderate and severe kidney insufficiency
* hepatic insufficiency
* history of hypercortisolism or adrenal insufficiency
* treatment interfering with the cortisol metabolism: taking oral or inhaled glucocorticoids within the last 6 months
* pregnant and lactating woman.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients suffering from FPL2 with the R482 codon mutation of the LMNA gene treated in the department of endocrinology at Lille University Hospital.
Sampling Method: Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2022-04-19 (Actual); Primary Completion 2023-11-09 (Actual); Study Completion 2023-11-09 (Actual)

PRIMARY OUTCOMES:
THE/(THF+αTHF) ratio measured in the 24h urine collections in patients | Baseline

SECONDARY OUTCOMES:
11BHSD1 expression in subcutaneous adipose tissue in patients | Baseline
Cortisol metabolites excretion in patients | Baseline
Correlation of 11BHSD1 activity and metabolic parameters in patients | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Stéphanie ESPIARD, MD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hop Claude Huriez, Lille, France